CLINICAL TRIAL: NCT04857749
Title: The Effects of Navigation in the Management of Symptoms Related to Head and Neck Radiotherapy: A Single Center Randomized Controlled Experimental Study
Brief Title: Navigation on Head and Neck Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ülkü Saygılı, Phd Student, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: USaygili1
Record Dates: First submitted 2021-04-17; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy; Navigation nursing; Symptom management; Quality of life; Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Data from patients in the control group will be collected as in the experimental group. In the first interview, the patients in the control group will be given a training booklet. Apart from this, the standard approach, treatment and care of the clinic will be applied to all patients.
  Interventions: Other: Standard care
- Navigation grup (Experimental): While the standard treatment approaches of the hospital are applied to all patients, a nursing navigation program will be applied in addition to the patients in the experimental group. The navigation program will be started on the first day of radiotherapy by giving a 30-minute visual training and handbook related to expected side effects. Afterwards, patient follow-up will continue with phone reminders and weekly follow-up for seven weeks.
  Interventions: Other: Navigation Nursing

INTERVENTIONS:
Other: Standard care — As a pre-test to the patients in the group just before starting treatment; Informed Consent Form, Patient Identification Form, CTCAE v5.0 toxicity criteria, Quality of Life Scale will be applied. At the end of the seven weeks, the post-test (measurement tools included in the pre-test) will be applied.
  Other Names: Follow-up
  Arms: Control group
Other: Navigation Nursing — With the role of navigator, the nurse contributes to increase the quality of care and to positively affect the physical, psychological and social well-being of the patient. Navigator nurses address patient barriers to care that are complex and often not easily resolved. As a result of the navigation nurses participating in care in the field of oncology; Providing assistance to the side effects of cancer and its treatment, including symptom preventive measures, supporting communication between individuals participating in treatment, preventing delays in treatment, explaining the language of medical treatment, providing psychosocial support, defining and recommending resources.
  Arms: Navigation grup

SUMMARY:
The aim of this experimental study is to evaluate the effect of nurse navigation in the management of symptoms associated with head and neck radiotherapy. All head and neck cancer patients who meet the study criteria of the Radiation Oncology Clinic of Selçuk University Medical Faculty Hospital will be included in the study. According to the previously prepared randomization list, the study group consisted of a total of 88 people, 41 in the experimental group and 47 in the control group. While the standard treatment approaches of the hospital are applied to all patients, a nursing navigation program will be applied in addition to the patients in the experimental group.Quality of life and toxicity criteria will be applied to all patients as measurement tools.

DETAILED DESCRIPTION:
The navigation program will be started on the day patients start their treatment. Before starting radiotherapy on the first day of radiotherapy, patients will be given a visual education guide about the radiotherapy treatment and the expected side effects. Afterwards, there will be a weekly follow-up with phone reminders. Inclusion criteria in the study; Being over the age of 18, the patient whose treatment and follow-up will continue for 7 weeks, patient diagnosed with head and neck cancer, scheduled to receive radiotherapy, patients who verbally and in writing approved to participate in the study after the explanation about the research. Exclusion criteria from the study; Metastasis development in the patient, refusing to participate in the research after the explanation about the research, the patient himself / herself wants to leave the study.For all patients included in the study, informed consent forms will be obtained just before starting treatment, and the patient identification form, CTCAE v5.0 toxicity criteria and EORTC QLQ-H & N35 scales will be applied. Quality of life measurements will be repeated at the end and middle of the treatment. In addition, weight measurements and laboratory follow-up of the patients will be done at the beginning and at the end of the study. NCSS (Number Cruncher Statistical System) 2007 program will be used for statistical analysis. Descriptive statistics, parametric and non-parametric tests will be used to evaluate data.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Being over the age of 18
* The patient whose treatment and follow-up will continue for 7 weeks
* Patient diagnosed with head and neck cancer, scheduled to receive radiotherapy
* Patients who verbally and in writing approved to participate in the study after the explanation about the research

Exclusion Criteria:

* Metastasis development in the patient
* Refusing to participate in the research after the explanation about the research.
* The patient himself / herself wants to leave the study.
* Treatment interruption for more than 2 days due to deterioration of the general condition of the patient
* Taking the patient into intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2021-06-20 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
CTCAE v5.0 Toxicity Criteria | 10 minute
  Mucositis, Dry mouth, Pain in the mouth, Dysphagia, Nausea, Constipation will be evaluated using the toxicity Criteria grading system. Grading is made as Grade 0,1,2,3,4.
EORTC QLQ C-30 | 12 minute
  It is applied to diagnose the quality of life of patients and the quality of life of individuals diagnosed with cancer. It is 30 questions in total. Likert type questions; Evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
EORTC QLQ-HN35 | 14 minute
  It is applied to diagnose the quality of life of patients with head and neck cancer and the quality of life of individuals diagnosed with cancer. It is 35 questions in total. Likert type questions; Evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
Patient Identification Form: | 10 minute
  Question form prepared by the researcher in line with the literature; It consists of a total of 26 questions with 17 open-ended and 9 closed-ended questions to evaluate the sociodemographic characteristics, disease-related characteristics and disease treatment characteristics of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duzova US, Can G. The effect of navigation programme on the management of symptoms related to head and neck radiotherapy. Transpl Immunol. 2021 Dec;69:101488. doi: 10.1016/j.trim.2021.101488. Epub 2021 Oct 20. PMID 34687909